CLINICAL TRIAL: NCT02155595
Title: Pathogenesis of Atypical Femur Fractures on Long Term Bisphosphonate Therapy
Acronym: NIH fracture
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Sudhaker D Rao, MD, Senior staff physician, Henry Ford Health System
Other Study IDs: 1R01AR062103-01A1 (NIH)
Record Dates: First submitted 2014-01-29; First posted 2014-06-04 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Osteoporosis; Atypical Femoral Fractures; Prodromal Bone Deterioration
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone & serum to be retained per institutional guidelines and clinical practice
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 500 with BP treatment: patients will undergo lab tests, X-ray, bone scan or MRI, as needed (90 of these individuals can opt for iliac crest bone biopsy)
  Interventions: Other: 500 with BP treatment
- 500 without BP treatment: patients will undergo lab tests, X-ray, bone scan or MRI, as needed
  Interventions: Other: 500 without BP treatment

INTERVENTIONS:
Other: 500 without BP treatment — lab tests, X-ray, bone scan or MRI, as needed
  Groups: 500 without BP treatment
Other: 500 with BP treatment — lab tests, X-ray, bone scan or MRI, as needed (90 of these individuals can opt for iliac crest bone biopsy)
  Groups: 500 with BP treatment

SUMMARY:
The purpose of this protocol is to determine the risk of atypical femoral shaft (thigh bone) fractures after long term fracture prevention therapy with a class of drugs called "bisphosphonates", colloquially referred to as Alendronate, risedronate, Ibandronate, and Zoledronate.

In addition, the study is designed to find out which patient is most likely to develop this potential life changing complication and why. Finally, the results of this study will help clinicians to better understand the reason and thus tailor patient specific treatments…i.e., "the right treatment for the right patient for right duration."

ELIGIBILITY:
Inclusion Criteria:

* women with a diagnosis of osteopenia or osteoporosis as defined by Bone Mineral density (BMD)
* patient treated with BPs for >5 years
* patients treated with non-BP anti-fracture medications such as...
* estrogens, raloxifene, calcitonin
* treatment naive patients

Exclusion Criteria:

* all men regardless of BMD result
* patients with obvious traumatic AFF
* patients with normal BMD (better than -1.0 T-score at spine or proximal hip)
* unable to take tetracycline
* previous use of teriparatide
* known allergies to the following:
* tetracycline antibiotics
* meperidine
* midazolam

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be found within the Henry Ford Health System Division of Endocrinology, Diabetes, Bone & Mineral Disorders
Sampling Method: Non-Probability Sample
Enrollment: 738 (Actual)
Dates: Start 2014-05; Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Prodromal bone deterioration (PBD) | 5 years
  Determine the prevalence of PBD and/or Atypical Femoral Fractures (AFF) in patients with post-menopausal or glucocorticoid related osteoporosis, either treated with bisphosphonate (BP) for more than 2 years or never treated with a BP

SECONDARY OUTCOMES:
Diagnosis of PBD | 5 years
  Refine diagnostic criteria for the diagnosis of PBD

OTHER OUTCOMES:
Osteocyte lacunae | 5 years
  Determine the prevalence of osteocyte lacunae. In BP treated patients with Severely Suppressed Bone Turnover (SSBT), PBD, or AFF, or with none of these complications, determine the prevalence of osteocyte lacunae in osteonal and interstitial iliac cortical bone

CONTACTS AND LOCATIONS:
Overall Officials: Sudhaker D. Rao, M.B;B.S., Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Medical Center, New Center One, Detroit, Michigan, United States

REFERENCES:
- [Derived] Farlay D, Rizzo S, Ste-Marie LG, Michou L, Morin SN, Qiu S, Chavassieux P, Chapurlat RD, Rao SD, Brown JP, Boivin G. Duration-Dependent Increase of Human Bone Matrix Mineralization in Long-Term Bisphosphonate Users with Atypical Femur Fracture. J Bone Miner Res. 2021 Jun;36(6):1031-1041. doi: 10.1002/jbmr.4244. Epub 2021 Feb 11. PMID 33434290